CLINICAL TRIAL: NCT00021073
Title: Phase I Study of Flavopiridol in Combination With 5-Fluorouracil, Leucovorin and Irinotecan in Patients With Advanced Malignancies
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02389; NCI-2012-02389 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000068745; MAYO-MC0014; NCI-2450; MC0014 (Other: Mayo Clinic); 2450 (Other: CTEP)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — alvocidib; Leucovorin; Fluorouracil; Irinotecan

ARMS (1):
- Treatment (alvocidib, combination chemotherapy) (Experimental): Group I: Patients receive FLAVO IV over 24 hours on day 1 and CF IV and 5-FU IV over 1.5 hours daily on days 2-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of FLAVO and 5-FU until the MTD are determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity.
  Once the MTDs for FLAVO and 5-FU are determined, patients receive FLAVO, CF, and 5-FU as in group I plus irinotecan IV over 1.5 hours on day 1. Courses repeat as in group I. Cohorts of 3-6 patients receive escalating doses of irinotecan until the MTD is determined. The MTD is defined as in group I.
  Interventions: Drug: alvocidib; Drug: leucovorin calcium; Drug: fluorouracil; Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E

SUMMARY:
Phase I trial to study the effectiveness of combining flavopiridol, fluorouracil, and leucovorin with or without irinotecan in treating patients who have advanced cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of flavopiridol, fluorouracil, and leucovorin calcium with or without irinotecan in patients with advanced malignancy.

II. Assess the toxic effects of these regimens in these patients. III. Determine the clinical response in patients treated with these regimens.

OUTLINE: This a dose-escalation study of flavopiridol (FLAVO), fluorouracil (5-FU), and irinotecan. Patients are assigned to 1 of 2 groups. Groups I and II are conducted sequentially.

Group I: Patients receive FLAVO IV over 24 hours on day 1 and leucovorin calcium (CF) IV and 5-FU IV over 1.5 hours daily on days 2-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of FLAVO and 5-FU until the maximum tolerated doses (MTD) are determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity.

Group II: Once the MTDs for FLAVO and 5-FU are determined, patients receive FLAVO, CF, and 5-FU as in group I plus irinotecan IV over 1.5 hours on day 1. Courses repeat as in group I. Cohorts of 3-6 patients receive escalating doses of irinotecan until the MTD is determined. The MTD is defined as in group I.

Patients are followed at 3 months.

PROJECTED ACCRUAL: A maximum of 57-90 patients will be accrued for this study within 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy

  * Unresectable tumor
  * No known standard therapy with curative potential or capability of extending life expectancy
* No untreated CNS metastases
* Performance status - ECOG 0-2
* At least 12 weeks
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 8 g/dL
* Direct bilirubin no greater than upper limit of normal (ULN)
* AST no greater than 3 times ULN (5 times ULN if liver metastases present)
* Creatinine no greater than 1.5 times ULN
* No New York Heart Association class III or IV heart disease
* No seizure disorder
* No uncontrolled infection
* No baseline diarrhea, defined as at least 4 loose or liquid stools/day
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* More than 4 weeks since prior biologic therapy
* More than 4 weeks since prior immunotherapy
* No concurrent immunotherapy
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and fully recovered from acute reversible effects
* No other concurrent chemotherapy
* More than 4 weeks since prior radiotherapy
* No prior radiotherapy to more than 25% of bone marrow
* No concurrent radiotherapy
* No other concurrent ancillary investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2001-05; Primary Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Number and severity of toxicity incidents of alvocidib, 5-fluorouracil, leucovorin calcium with and without irinotecan hydrochloride, graded according to the National Cancer Institute Common Toxicity Criteria (NCI CTC) v2.0 | Up to 5 years

SECONDARY OUTCOMES:
Number of responses (complete response, partial response, stable disease, and progressive disease) assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 5 years
  Summarized by simple descriptive summary statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Bible, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States